CLINICAL TRIAL: NCT06916312
Title: Airways to Alteration: Investigating the Impact of Breathwork & Meditation on Conscious State
Brief Title: Comparing Effects of Intense Breathwork to Meditation on Altered States of Consciousness
Acronym: A2A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sussex (Other)
Collaborators: DMT Quest (Unknown); ResearchHub (Unknown)
Responsible Party: Principal Investigator, Guy Fincham, PhD, University of Sussex
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ER/GF221/9
Record Dates: First submitted 2025-03-24; First posted 2025-04-08 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Altered States of Consciousness; Wellbeing
Keywords: Breathwork
MeSH Terms: interventions — Meditation; Whole Body Imaging

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditation (Active Comparator): Single guided body scan meditation session.
  Interventions: Behavioral: Meditation
- High ventilation breathwork (Experimental): Single guided conscious connected breathing session.
  Interventions: Behavioral: High ventilation breathwork

INTERVENTIONS:
Behavioral: High ventilation breathwork — Single guided conscious connected breathing session.
  Other Names: Conscious connected breathing
  Arms: High ventilation breathwork
Behavioral: Meditation — Single guided body scan meditation session.
  Other Names: Body scan
  Arms: Meditation

SUMMARY:
This study aims to investigate the impact of high ventilation breathwork (HVB) and meditation on altered states of consciousness (ASCs). The study will compare the effects of a single guided HVB session to a single guided body scan meditation session. The primary aim is to explore the impact of HVB and meditation on ASCs, while secondary aims relate to mental health and wellbeing.

DETAILED DESCRIPTION:
The study is a randomised controlled trial (RCT) involving up to 24 healthy adult participants who have prior experience with HVB. Participants will be randomly allocated to either the HVB or meditation group. The study will assess outcomes such as altered states of consciousness, mystical experiences, emotional breakthroughs, and overall wellbeing.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults in Brighton and the surrounding area
* Prior experience practising high ventilation breathwork in the form of conscious connected breathing
* No history of adverse events during such prior breathwork sessions.

Exclusion Criteria:

* History of hypotension
* Hypertension
* Respiratory or cardiovascular problems
* Fainting or syncope
* Epilepsy or seizures
* Panic disorder or panic attacks
* Cerebral aneurysm
* Pregnancy (and possibility one might be pregnant, trying to get pregnant, or are breastfeeding)
* Breathlessness
* Bradypnea
* Tachypnoea
* Any mental/physical issues affecting the ability to engage in breath control activities.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-06-16 (Actual)

PRIMARY OUTCOMES:
Altered states of consciousness | Immediately after the intervention.
  Five Dimensions of Altered States of Consciousness Scale. Comprises five subscales: oceanic boundlessness, dread of ego dissolution, visionary restructuralisation, auditory alterations and vigilance reduction. Scores range from 0 to 100, with higher scores indicating more profound altered states of consciousness.
Mystical experience | Immediately after the intervention.
  Mystical Experience Questionnaire Brief. Comprises four subscales: transcendence, positive mood, ineffability, and mystical. Scores range from 0 to 20, with higher scores indicating a more profound mystical experience.
Emotional breakthrough | Immediately after the intervention.
  Emotional Breakthrough Inventory. Scores range from 0 to 100, with higher scores indicating greater levels of emotional breakthrough (reflecting a better outcome).

SECONDARY OUTCOMES:
Psychological insight | Post-intervention (one week after the intervention).
  Psychological Insight Scale. Scores range from 0 to 100, with higher scores indicating greater psychological insight. An additional item separately evaluates self-reported behavioural change resulting from a psychedelic experience.
Depersonalisation | Immediately after the intervention.
  Cambridge Depersonalisation Scale (State-Version). Scores range from 0 to 100, with higher scores indicating greater levels of dissociative symptoms.
Fatigue | Baseline and post-intervention (one week before and after the intervention).
  Shortened Fatigue Questionnaire. Scores range from 4 to 28, with higher scores indicating more severe fatigue.
Sleep-related impairment | Baseline and post-intervention (one week before and after the intervention).
  PROMIS Item Bank v. 1.0 - Sleep-Related Impairment - Short Form 4a (score range: 5-20; higher scores denote worse outcome). Data scored using a T-score transformation according to PROMIS Sleep scoring manual on: www.healthmeasures.net
Mental wellbeing | Baseline and post-intervention (one week before and after the intervention).
  Short Warwick-Edinburgh Mental Wellbeing Scale (SWEMWBS) (score range: 7 to 35; higher scores denote better outcome). Total raw scores are then transformed into metric scores using the SWEMWBS conversion table on: www.warwick.ac.uk
Depressive symptoms, anxiety, and stress | Baseline and post-intervention (one week before and after the intervention).
  Depression Anxiety Stress Scale-21 (DASS-21) - stress, anxiety and depression subscales (score range for each: 0-21; higher scores denote worse outcomes). Score on DASS-21 then multiplied by two to convert it to the longer form DASS-42 final score.

OTHER OUTCOMES:
Psychedelic experience predictiveness | After completing consent form to participate in the study.
  Imperial Psychedelic Predictor Scale. Scores range from 0 to 100, with higher scores donating higher predictiveness of having a psychedelic experience. Additional items assess rapport.
General experience | One week post-intervention.
  Open-ended, free text.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sussex, Brighton, Sussex, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-09): https://cdn.clinicaltrials.gov/large-docs/12/NCT06916312/Prot_SAP_000.pdf